CLINICAL TRIAL: NCT05969678
Title: Effects of Respiratory Training Intervention on Lung Capacity and Quality of Life of Community Elderly
Brief Title: Respiratory Training Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chung Shan Medical University (Other)
Responsible Party: Principal Investigator, Hsiang Chu Pai, Principal Investigator, Chung Shan Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 202304111RINC
Record Dates: First submitted 2023-07-23; First posted 2023-08-01 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Elders
Keywords: breathing training; abdominal diaphragmatic breathing; respiratory capacity; Quality of Life-
MeSH Terms: interventions — Breathing Exercises

STUDY DESIGN:
Intervention Model Description: The experimental group will receive the breathing training of abdominal diaphragmatic breathing method combined with incentive spiromete. The control group is only taught the breathing training of abdominal diaphragmatic breathing.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group ( breathing training with incentive spiromete) (Experimental): The experimental group will receive the breathing training of abdominal diaphragmatic breathing method combined with incentive spiromete.
  Interventions: Behavioral: breathing training
- control group (No Intervention): The control group is only taught the breathing training of abdominal diaphragmatic breathing.

INTERVENTIONS:
Behavioral: breathing training — receive the breathing training of abdominal diaphragmatic breathing method combined with incentive spiromete
  Arms: Intervention group ( breathing training with incentive spiromete)

SUMMARY:
This study aims to examine the effect of abdominal diaphragmatic breathing combined with incentive spirometer breathing training on the lung capacity of elderly community residents.

DETAILED DESCRIPTION:
The research will be conducted in a community in central Taiwan. Inclusion criteria are people over the age of 65 in the community. All participants will be randomly assigned to either the experimental group or the control group. The experimental group will receive the breathing training of abdominal diaphragmatic breathing method combined with incentive spiromete. The control group is only taught the breathing training of abdominal diaphragmatic breathing. Four assessment tools will be used, including the demographic questionnaire, respiratory capacity indicators, Modified Medical Research Council (mMRC) Dyspnea Scale, and the World Health Organization Quality of Life-BREF Taiwan Version (WHOQOL-BREF; WHOQOL-BREF). Data analysis will be performed by independent sample t test, paired t test, and repeated measures analysis. All data analysis will be performed by SPSS version 22.0.

ELIGIBILITY:
Inclusion Criteria:

1. Over 65 years old
2. A person who is conscious and can communicate in Mandarin or Hokkien, and can cooperate with breathing exercises.
3. Agree to interview or fill out the questionnaire, and complete the consent form.

Exclusion Criteria:

1. Hemoptysis, pneumothorax, unstable cardiovascular status, chronic respiratory diseases (asthma, chronic obstructive pulmonary disease).
2. Recent myocardial infarction or pulmonary embolism, thoracic aortic aneurysm, abdominal aortic aneurysm or cerebral aneurysm, recent eye surgery, nausea or vomiting, recent chest or abdominal surgery.
3. Suffering from infectious diseases: airborne such as: chickenpox, measles, tuberculosis, severe special infectious pneumonia influenza. Droplet transmission such as: pneumonia, influenza.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 128 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2023-08-10 (Actual); Study Completion 2023-12-08 (Actual)

PRIMARY OUTCOMES:
respiratory capacity indicators | The questionnaire will be filled 3 times, during the first and fourth, and eighth weeks of the study.
  Indicator: FVC (forced vital capacity) ,FEV1(forced expiratory volume),MVV (maximal voluntary ventilation).
Dyspnea | The questionnaire will be filled 3 times, during the first and fourth, and eighth weeks of the study.
  Modified Medical Research Council (mMRC) Dyspnea Scale) will be used to assess participants' breathing condition. This scale consisting of five items containing statements about the impact of breathlessness on the individual . It ranges from grade 0 to 4. Higher scores reflect lower respiratory function condition.
Quality of Life (OL) | The questionnaire will be filled 3 times, during the first and fourth, and eighth weeks of the study.
  The 28 items World Health Organization Quality of Life-BREF Taiwan Version (WHOQOL-BREF)WHOQOL-BREF) will be used to examine participants' quality of life. Each item is rated on a 5-point Likert-type scale ranging from 1 (not at all) to 4 (very agree). The total score is the sum of all item scores. Higher scores reflect greater quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Hsiang Chu Pai, PhD, Study Director — Chung Shan Medical University
Locations (1):
- Chung Shan Medical University, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No